CLINICAL TRIAL: NCT04035148
Title: Cardiopulmonary Exercise Test in Evaluation of Pulmonary Hypertension in COPD Patients
Brief Title: CPET in Evaluation of PH in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Emad El-din Abdalah, Principal investigator, Assiut University
Other Study IDs: CPET in PH in COPD
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: COPD; Pulmonary Hypertension Secondary
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test; Echocardiography; Respiratory Function Tests; Blood Gas Analysis; Electrocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test — we prepared incremental treadmill exercise protocol in which the work rate increased at one-minute intervals.Transthoracic Echocardiography(TTE) : The first step non-invasive method to diagnose PHT.
  Other Names: Echocardiography; pulmonary function test; blood gases; Electrocardiography

SUMMARY:
* To evaluate the entire course of exercise during CPET in COPD patients.
* To study whether CPET, PFTs and arterial blood gases could discriminate between COPD patients with and without PH.
* To study whether the existence of pulmonary hypertension in COPD is related to characteristic findings in gas exchange and circulatory parameters during cardiopulmonary exercise testing (CPET).

DETAILED DESCRIPTION:
(COPD) is a common cause of pre-capillary pulmonary hypertension (PH). Pulmonary hypertension (PHT) is a common complication of COPD and is determinant for the prognosis of COPD.

PHT is defined as A mean PAP of ≥ 25 mmHg measured by right heart catheterization at rest.

Exercise tolerance in patients with COPD is reduced due to ventilatory limitation, gas exchange abnormalities, and deconditioning as the disease progresses, and this may impair functional capacity and the quality of life.

COPD patients usually terminate physical activity when the ventilatory requirement exceeds their maximal ventilatory capacity.

If they have PH, the altered hemodynamic response may reduce their exercise capacity further.

Nowadays, despite the fact that LTOT improves the survival of hypoxaemic patients, PH is still associated with lower survival rates . Importantly, an elevated Ppa was also associated with an increased risk of severe acute exacerbation in COPD patients with moderate-to-severe airflow limitation .

Impaired exercise tolerance in COPD patients would suggest that cardiopulmonary exercise test (CPET) is a valuable tool to reveal whether they have PH or not.

Transthoracic echocardiography (TTE) is one such tool and is widely available and safe. In addition to its role in diagnosis, it can be used to screen for high-risk patient populations, to assess prognosis and to monitor disease stability and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD patients
* with age ≥ 40 years.
* Prior to inclusion, the COPD diagnosis was verified by spirometry before and after bronchodilation.
* treatment was optimized and Patients on regular medication.

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Patients underwent thorough pulmonary and cardiologic preinclusion screening, and those with pulmonary disease other than COPD and emphysema.
* arrhythmia
* valvular or coronary heart disease
* left ventricle dysfunction
* obstructive sleep apnea syndrome
* pulmonary embolism
* systemic hypertension ≥160/90 mmHg
* inflammatory disease
* hyperthyroidism
* renal failure
* inability to exercise (due to orthopedic, neurologic or musculoskeletal problem).

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stable chronic obstructive pulmonary disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of oxygen uptake during cardiopulmonary exercise testing (% predicted) | Baseline
  For the assessment whether the existence of pulmonary hypertension in COPD is related to characteristic findings during cardiopulmonary exercise testing (CPET).
Measurement the arterial pO2 in mmHg and arterial pCO2 at baseline | Baseline
  The blood gases pO2 and pCO2 are taken to characterize the gas exchange during cardiopulmonary exercise which is a routine procedure

SECONDARY OUTCOMES:
measurement of symptoms quantified by COPD Assessment Test (CAT Assessment)- total score 40. | Baseline
  For the assessment of the symptoms of the study group and its relation to exercise capacity and the impact COPD on wellbeing and daily life - CAT score < 10 is associated with better outcome and prognosis but score = or > 10 is associated with poor outcome and prognosis.
measurement of dyspnoea quantified by the modified Medical Research Council (mMRC) Dyspnea Scale (grades from 0 to 4 ) | Baseline
  measures perceived respiratory disability indicating the extent to which their breathlessness affects their mobility - dyspnoea is assessed by accepted questionnaires typically used for COPD patients at baseline- grade <2 indicates better outcome and prognosis but grade = or >2 indicates poor outcome and prognosis.
Measurement of FEV1 | Baseline
  For assessment of which degrees of severity of COPD are more related to development of COPD with pulmonary hypertension.
Measurement of Breathing reserve during cardiopulmonary exercise testing | Baseline
  The breathing reserve in % is assessed at the end of the cardiopulmonary exercise testing to characterize a ventilatory limitation of the exercise test. It is calculated as percent from the minute ventilation in relation to the maximum mandatory ventilation. The measurement is a routine measurement during cardiopulmonary exercise testing.
Measurement of Oxygen pulse during cardiopulmonary exercise testing | Baseline
Presence of cardiovascular comorbidities | Baseline
  For the cardiopulmonary characterization clinical characteristics, lung function, blood gases, laboratory investigation, ECG and echocardiography were used in addition to cardiopulmonary exercise testing.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Skjorten I, Hilde JM, Melsom MN, Hisdal J, Hansteen V, Steine K, Humerfelt S. Cardiopulmonary exercise test and PaO2 in evaluation of pulmonary hypertension in COPD. Int J Chron Obstruct Pulmon Dis. 2017 Dec 22;13:91-100. doi: 10.2147/COPD.S150034. eCollection 2018. PMID 29339921
- [Background] Sarac R, Cikes I, Butkovic D, Dimov-Butkovic D. [Doppler echocardiography in the evaluation of pulmonary hypertension in chronic obstructive pulmonary disease]. Lijec Vjesn. 1995 Jan-Feb;117(1-2):9-15. Croatian. PMID 7651072
- [Background] Habib G, Torbicki A. The role of echocardiography in the diagnosis and management of patients with pulmonary hypertension. Eur Respir Rev. 2010 Dec;19(118):288-99. doi: 10.1183/09059180.00008110. PMID 21119187
- [Background] Holverda S, Bogaard HJ, Groepenhoff H, Postmus PE, Boonstra A, Vonk-Noordegraaf A. Cardiopulmonary exercise test characteristics in patients with chronic obstructive pulmonary disease and associated pulmonary hypertension. Respiration. 2008;76(2):160-7. doi: 10.1159/000110207. Epub 2007 Oct 25. PMID 17960052
- See also: Holverda S et al. Respiration. (2008) — http://www.ncbi.nlm.nih.gov/pubmed/?term=Cardiopulmonary+exercise+test+characteristics+in+patients+with+chronic+obstructive+pulmonary+disease+and+associated+pulmonary+hypertension